CLINICAL TRIAL: NCT05838989
Title: Randomized Controlled Trial Comparing the Effectiveness of Stretching and Orthoses Versus Orthoses Alone in Individuals With Carpal Tunnel Syndrome
Brief Title: The Effectiveness of Stretching and Orthoses in Individuals With Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy ElMeligie, Lecturer of Physical Therapy and Director of Electromyography Lab, Ahram Canadian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012/0701
Record Dates: First submitted 2023-04-20; First posted 2023-05-03 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into one of three groups: stretching and prefabricated orthoses, orthoses alone, or a placebo treatment.
Who Masked: Outcomes Assessor
Masking Description: Participants and care providers will not be blinded to the treatment group, but outcomes assessors will be blinded to the treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: Stretching and Prefabricated Orthoses (Experimental): Participants in this arm will receive supervised general and lumbrical muscle stretching exercises for 10 minutes, three times per week, for 8 weeks, as well as prefabricated wrist orthoses.
  Interventions: Device: Prefabricated Orthoses; Other: general and lumbrical muscle stretching
- Group B: Orthoses Alone (Experimental): Participants in this arm will receive prefabricated wrist orthoses only.
  Interventions: Device: Prefabricated Orthoses
- Group C: Placebo Treatment (Placebo Comparator): Participants in this arm will receive placebo treatment consisting of gentle wrist and hand movements.
  Interventions: Other: Placebo

INTERVENTIONS:
Device: Prefabricated Orthoses — Participants in this group will be provided with prefabricated wrist orthoses to wear during the day and at night to provide support and immobilization to the wrist. Participants will be instructed to wear the orthoses as directed by their healthcare provider.
  Arms: Group A: Stretching and Prefabricated Orthoses; Group B: Orthoses Alone
Other: general and lumbrical muscle stretching — Participants in this group will receive supervised general and lumbrical muscle stretching exercises for 10 minutes, three times per week, for 8 weeks. The stretching exercises will be performed under the supervision of a trained therapist and will include a series of exercises designed to stretch the muscles in the hands, wrists, and forearms. In addition, participants will be provided with prefabricated wrist orthoses to wear during the day and at night to provide support and immobilization to the wrist.
  Arms: Group A: Stretching and Prefabricated Orthoses
Other: Placebo — Participants in this group will receive placebo treatment consisting of gentle wrist and hand movements. The movements will be performed under the supervision of a trained therapist and will consist of gentle range of motion exercises designed to mobilize the joints in the hands and wrists. Participants will not be provided with any orthoses to wear during the study.
  Arms: Group C: Placebo Treatment

SUMMARY:
The objective of this study is to compare the effectiveness of stretching and prefabricated orthoses versus orthoses alone in individuals with carpal tunnel syndrome (CTS) using validated condition-appropriate outcome measures such as BCTQ, pain levels, grip strength, and nerve conduction studies.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 30-60 years or older with a confirmed diagnosis of carpal tunnel syndrome based on clinical presentation and/or nerve conduction studies.
2. Participants must have a moderate level of symptom severity, defined as a score of 2 or greater on the symptom severity subscale of the Boston Carpal Tunnel Questionnaire (BCTQ).
3. Participants must have a moderate level of functional impairment, defined as a score of 2 or greater on the functional status subscale of the BCTQ.
4. Participants must be willing and able to provide informed consent to participate in the study.

Exclusion Criteria:

1. Participants with a history of hand or wrist surgery within the past 6 months, as this could impact hand function and confound the study results.
2. Participants with severe hand or wrist pain that would prevent completion of the outcome measures or interfere with their ability to participate in the study.
3. Participants with severe cognitive impairment or language barrier that would prevent understanding of the study instructions or interfere with their ability to participate in the study.
4. Participants with any other medical condition that could affect hand function or interfere with test completion, such as rheumatoid arthritis, osteoarthritis, or peripheral neuropathy.
5. Participants who have participated in any other clinical trial or research study involving the hand or wrist within the past 3 months, as this could impact hand function and confound the study results.
6. Participants who are unable to comply with study procedures or follow-up requirements, such as attending scheduled study visits or completing study questionnaires.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Boston Carpal Tunnel Questionnaire (BCTQ) | Changes in BCTQ at baseline, 8 weeks, and 16 weeks.
  The BCTQ is a validated condition-specific questionnaire used to assess the severity of symptoms and functional limitations associated with carpal tunnel syndrome. The questionnaire consists of 11 items related to symptom severity and 8 items related to functional status. The scores for each set of items are combined to generate symptom severity and functional status scores, which will be used as the primary outcome measures for this study.
Pain Levels | Changes in pain level at baseline, 8 weeks, and 16 weeks.
  Pain levels will be assessed using a visual analogue scale (VAS) ranging from 0 (no pain) to 10 (worst pain imaginable). Participants will be asked to rate their pain levels at rest and during specific activities such as gripping, pinching, and typing.

SECONDARY OUTCOMES:
Grip Strength | Changes in grip strength at baseline, 8 weeks, and 16 weeks.
  Grip strength will be measured using a hand-held dynamometer. Participants will be instructed to grip the dynamometer as hard as possible, and the maximum force generated will be recorded in kilograms. Grip strength is a commonly used outcome measure in hand rehabilitation research and is a reliable and valid measure of hand function.
Nerve Conduction Studies | Changes in nerve conduction studies at baseline, 8 weeks, and 16 weeks.
  Nerve conduction studies will be used to assess the severity and extent of median nerve involvement in participants with carpal tunnel syndrome. The studies will be performed by a trained neurophysiologist using standard techniques and equipment.

CONTACTS AND LOCATIONS:
Overall Officials: Amal Fawzy, Ph.d, Study Chair — Faculty of Physical Therapy, Ahram Canadian University
Locations (1):
- Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data (IPD) collected during this study will be available upon reasonable request. Requests for access to the data should be submitted via email to mohamed.elmeligie@acu.edu.eg. All requests will be reviewed by the study investigators to ensure that they are reasonable and consistent with the ethical principles of the study. Access to the data will be granted in compliance with applicable laws and regulations, and with appropriate safeguards to protect the privacy and confidentiality of study participants.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: During the trial and 1 year after it ends
Access Criteria: via email to mohamed.elmeligie@acu.edu.eg